CLINICAL TRIAL: NCT04328259
Title: Prevalance of non_ Alcoholic Fatty Liver Diseases in Patient With Inflammatory Bowel Diseases Attending Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Al shymaa aAdel hakm Ahmed Ali, Principal Investigator, Assiut University
Other Study IDs: NAFLD in patient of IBD
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Disease Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
To assess the prevalance of non_alcoholic fatty liver diseases in inflammatory bowel disease patients and its relation to type of treatment given and disease severity

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) including Crohns disease (CD) and ulcerative colitis (UC) are chronic relapsing disorders that often require long-term therapy and follow up .

They are recognized for their complex pathophysiology that involves innate immune system deregulation and altered microbiome in genetically predisposed individuals. Non-alcoholic fatty liver disease (NAFLD) includes a wide spectrum of disorders, ranging from hepatic steatosis (NAFL) to non-alcoholic steatohepatitis (NASH). NAFLD patients are at high risk for liver fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). Also NAFLD is typically associated with altered metabolism and metabolic syndrome (MetS).

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease (CD) patients
* ulcerative colitis (UC) patients

Exclusion Criteria:

* diabetic patients
* BMI equal and more than 30.0-34.9(class I obesity)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Inflammatory bowel disease patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
the prevalance of non-alcoholic fatty liver in inflammatory bowel disease participants | one year
  u/s will be done to all participants of inflammatory bowel disease to asses the rate of non-alcoholic fatty liver affection of all patients

SECONDARY OUTCOMES:
the Correlation between immunosuppressive drugs and prevalance of non-alcoholic fatty liver affection in inflammatory bowel disease participants | one year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torres J, Mehandru S, Colombel JF, Peyrin-Biroulet L. Crohn's disease. Lancet. 2017 Apr 29;389(10080):1741-1755. doi: 10.1016/S0140-6736(16)31711-1. Epub 2016 Dec 1. PMID 27914655
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] de Souza HS, Fiocchi C. Immunopathogenesis of IBD: current state of the art. Nat Rev Gastroenterol Hepatol. 2016 Jan;13(1):13-27. doi: 10.1038/nrgastro.2015.186. Epub 2015 Dec 2. PMID 26627550
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Demir M, Lang S, Steffen HM. Nonalcoholic fatty liver disease - current status and future directions. J Dig Dis. 2015 Oct;16(10):541-57. doi: 10.1111/1751-2980.12291. PMID 26406351
- [Background] Wong VW, Wong GL, Choi PC, Chan AW, Li MK, Chan HY, Chim AM, Yu J, Sung JJ, Chan HL. Disease progression of non-alcoholic fatty liver disease: a prospective study with paired liver biopsies at 3 years. Gut. 2010 Jul;59(7):969-74. doi: 10.1136/gut.2009.205088. PMID 20581244
- [Background] Calzadilla Bertot L, Adams LA. The Natural Course of Non-Alcoholic Fatty Liver Disease. Int J Mol Sci. 2016 May 20;17(5):774. doi: 10.3390/ijms17050774. PMID 27213358
- [Background] McPherson S, Hardy T, Henderson E, Burt AD, Day CP, Anstee QM. Evidence of NAFLD progression from steatosis to fibrosing-steatohepatitis using paired biopsies: implications for prognosis and clinical management. J Hepatol. 2015 May;62(5):1148-55. doi: 10.1016/j.jhep.2014.11.034. Epub 2014 Dec 1. PMID 25477264
- [Background] Gomollon F, Dignass A, Annese V, Tilg H, Van Assche G, Lindsay JO, Peyrin-Biroulet L, Cullen GJ, Daperno M, Kucharzik T, Rieder F, Almer S, Armuzzi A, Harbord M, Langhorst J, Sans M, Chowers Y, Fiorino G, Juillerat P, Mantzaris GJ, Rizzello F, Vavricka S, Gionchetti P; ECCO. 3rd European Evidence-based Consensus on the Diagnosis and Management of Crohn's Disease 2016: Part 1: Diagnosis and Medical Management. J Crohns Colitis. 2017 Jan;11(1):3-25. doi: 10.1093/ecco-jcc/jjw168. Epub 2016 Sep 22. PMID 27660341
- [Background] Magro F, Gionchetti P, Eliakim R, Ardizzone S, Armuzzi A, Barreiro-de Acosta M, Burisch J, Gecse KB, Hart AL, Hindryckx P, Langner C, Limdi JK, Pellino G, Zagorowicz E, Raine T, Harbord M, Rieder F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 1: Definitions, Diagnosis, Extra-intestinal Manifestations, Pregnancy, Cancer Surveillance, Surgery, and Ileo-anal Pouch Disorders. J Crohns Colitis. 2017 Jun 1;11(6):649-670. doi: 10.1093/ecco-jcc/jjx008. No abstract available. PMID 28158501
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Satsangi J, Silverberg MS, Vermeire S, Colombel JF. The Montreal classification of inflammatory bowel disease: controversies, consensus, and implications. Gut. 2006 Jun;55(6):749-53. doi: 10.1136/gut.2005.082909. PMID 16698746
- [Background] Saverymuttu SH, Joseph AE, Maxwell JD. Ultrasound scanning in the detection of hepatic fibrosis and steatosis. Br Med J (Clin Res Ed). 1986 Jan 4;292(6512):13-5. doi: 10.1136/bmj.292.6512.13. PMID 3080046
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702